CLINICAL TRIAL: NCT00494052
Title: An Intervention to Enhance CHD Risk Factor Modification: The Heart to Heart Feasibility Study
Brief Title: Evaluating a Web-Based Educational Program for Adults at Risk for Coronary Heart Disease (The Heart to Heart Feasibility Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Stacey Sheridan, MD, Stacey L. Sheridan, MD, MPH, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 490; K23HL074375-02 (NIH)
Record Dates: First submitted 2007-06-28; First posted 2007-06-29 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Coronary Disease; Cardiovascular Diseases
Keywords: Coronary Heart Disease; Choice Behavior; Risk Factors; Risk Assessment; Primary Prevention; Decision Making; Decision Aids; Patient Compliance
MeSH Terms: conditions — Coronary Disease; Cardiovascular Diseases; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Heart to Heart intervention
  Interventions: Behavioral: Heart to Heart (Web-Based Decision Aid); Behavioral: Physician Education Session
- 2 (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Heart to Heart (Web-Based Decision Aid) — Participants in the intervention group will access Heart to Heart, a Web site designed to educate them about their overall CHD risk, specific risk factors, and strategies and preferences for risk reduction.
  Arms: 1
Behavioral: Physician Education Session — A physician education session will be included in the program.
  Arms: 1

SUMMARY:
Coronary heart disease (CHD) is the leading cause of death in the United States, but fewer than half of all individuals at risk for CHD take advantage of proven strategies to lower their chances of developing this disease. This study will assess the effectiveness of Heart to Heart, a Web-based program, at educating people on ways to incorporate CHD risk-reduction strategies into their lives.

DETAILED DESCRIPTION:
CHD affects 13 million people in the United States. It is the leading cause of death in this country, and each year more than half a million Americans die from this disease. People who take steps to lower their cholesterol and blood pressure levels, lose weight, and stop smoking may be less likely to develop CHD. However, fewer than half of all individuals at risk for developing CHD follow these suggestions. Involving patients in the decision-making process regarding their medical care may improve their adherence to effective CHD prevention strategies. The goal of the Heart to Heart program is to provide information about CHD risk factors and encourage people to incorporate the appropriate risk-reduction measures into their lives. The purposes of this pilot study are to evaluate the ability of study researchers to recruit individuals with a moderate to high risk of CHD to participate in the study; to conduct a four-part CHD intervention (Heart to Heart) in a busy medical practice setting; and to measure participants' decision-making plans, self-reported adherence to medications, and changes in overall CHD risk factors. The results from this study will be used to guide future clinical trials.

This study will enroll patients being treated at the General Internal Medicine Clinic at the University of North Carolina at Chapel Hill who have a moderate to high risk of developing CHD. At an initial study visit, participants will complete questionnaires that assess CHD risk-reduction strategies, smoking status, and aspirin use. Blood pressure and cholesterol levels will also be measured. Participants will then be randomly assigned to either participate in the Heart to Heart intervention or receive usual care. Participants in the intervention group will access Heart to Heart, a Web site designed to educate them about their overall CHD risk, specific risk factors, and strategies and preferences for risk reduction. A Web-based coaching tool will encourage participants to talk with their doctor about risk-reduction choices. Participants will also receive brief adherence messages via the Web site 2, 4, and 6 weeks following their initial study visit. The messages will be designed to help participants adhere to their decisions. All participants will attend a study visit at Month 3 for repeat baseline testing. Following this visit, participants will receive a letter that includes their test results and their recalculated CHD risk. Participants may be contacted to take part in a focus group following the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Currently a patient at the General Internal Medicine Clinic at the University of North Carolina at Chapel Hill
* Moderate (6% to 20%) or high (greater than 20%) risk of CHD, as defined by current evidence and practice-based guidelines for aspirin use and cholesterol levels

Exclusion Criteria:

* Known cardiovascular disease (e.g., previous heart attack, previous coronary artery bypass graft or percutaneous coronary intervention, angina, previous transient ischemic attack [TIA] or stroke, peripheral vascular disease, congestive heart failure)
* Diabetes
* Low global risk of CHD (less than 6%)
* Dementia or other severe cognitive dysfunction
* Blindness
* Serious medical illness that would make the individual a poor candidate for the study (e.g., kidney failure, liver cirrhosis, HIV, non-skin cancer, any other illness for which their life expectancy is projected at less than 5 years)
* Inability to speak and understand English
* Participation in the preliminary study or in cognitive testing of intervention components

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2007-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of subject recruitment; feasibility of delivery of the CHD intervention and surveys in a busy practice setting; feasibility of measuring study outcomes | Measured at the end of the study period (approximately 2 years)

SECONDARY OUTCOMES:
Self-reported use of any new CHD risk reduction strategy; global CHD risk; blood pressure; serum total cholesterol and HDL-c levels; smoking status; aspirin use; self-reported plans for CHD risk reduction; self-efficacy for CHD risk reduction | Measured at participants' Month 3 study visit

CONTACTS AND LOCATIONS:
Overall Officials: Stacey L. Sheridan, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - UNC General Internal Medicine Clinic, Chapel Hill, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina

REFERENCES:
- [Background] Sheridan SL, Shadle J, Simpson RJ Jr, Pignone MP. The impact of a decision aid about heart disease prevention on patients' discussions with their doctor and their plans for prevention: a pilot randomized trial. BMC Health Serv Res. 2006 Sep 27;6:121. doi: 10.1186/1472-6963-6-121. PMID 17005051
- [Derived] Sheridan SL, Draeger LB, Pignone MP, Keyserling TC, Simpson RJ Jr, Rimer B, Bangdiwala SI, Cai J, Gizlice Z. A randomized trial of an intervention to improve use and adherence to effective coronary heart disease prevention strategies. BMC Health Serv Res. 2011 Dec 5;11:331. doi: 10.1186/1472-6963-11-331. PMID 22141447
- See also: Click here for the Heart to Heart Web site — http://www.med-decisions.com